CLINICAL TRIAL: NCT00587535
Title: Evaluation of a New MR Pulse Sequence to Quantify Liver Iron Concentration
Status: Completed | Type: Observational
Sponsor: Mayo Clinic (Other)
Responsible Party: Principal Investigator, Jeff Fidler, Professor of Radiology College of Medicine, Mayo Clinic
Other Study IDs: 1478-03
Record Dates: First submitted 2007-12-21; First posted 2008-01-07 (Estimated); Last update posted 2016-01-22 (Estimated); Status verified 2016-01

CONDITIONS: Hemochromatosis
Keywords: hemochromatosis; liver cirrhosis; liver diseases
MeSH Terms: conditions — Hemochromatosis; Liver Cirrhosis; Liver Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Hemochromatosis: Hemochromatosis
- Living-related liver donation: Living-related liver donation

SUMMARY:
The purpose of this study is to determine if a new MR pulse sequence is accurate in determining how much iron is in the liver.

DETAILED DESCRIPTION:
Quantification of liver iron requires liver biopsy and histological assessment. New rapid MR techniques allow determination of liver relaxation times that can be altered with increasing iron deposition. The purpose of this study is to compare the results obtained with MRI to liver biopsy and iron quantification in patients undergoing liver biopsy in the setting of hemochromatosis.

ELIGIBILITY:
Inclusion Criteria:

* Undergoing liver biopsy for suspected or known hemochromatosis
* Undergoing liver biopsy for living-related liver donation evaluation

Exclusion Criteria:

* Contraindication to MRI

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Gastroenterology Clinic; Liver Transplant Center; Surgery Clinic
Sampling Method: Non-Probability Sample
Enrollment: 18 (Actual)
Dates: Start 2003-08; Primary Completion 2011-07 (Actual); Study Completion 2011-07 (Actual)

PRIMARY OUTCOMES:
Accuracy of MR in quantifying liver iron | one time point

CONTACTS AND LOCATIONS:
Overall Officials: Jeff L Fidler, MD, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic, Rochester, Minnesota, United States

IPD SHARING:
Plan to Share IPD: No